CLINICAL TRIAL: NCT00153452
Title: Workplace Productivity of Persons Who Use Controlling Behavior With Intimate Partners
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Harvard University (Other)
Other Study IDs: CDC-NCIPC-4606
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: perpetration of intimate partner violence

SUMMARY:
The goal of this project is to pilot-test an instrument that is designed to assess the relationship between persons who use controlling behavior with intimate partners, as a risk factor for perpetrating intimate partner violence, and workplace productivity. The goal is to validate a survey instrument that can be applied to other workplace settings to measure productivity losses associated with controlling and aggressive behavior, which will serve to inform the development of workplace interventions designed to prevent intimate partner violence (IPV). This pilot-test will include two components of a survey conducted with employees in a workplace setting: questions to determine one's controlling behavior or propensity for violence in an intimate relationship, and questions designed to assess levels of productivity as measured by days missed from work (absenteeism) and days at work with diminished functional output (presenteeism). We expect productivity to decrease as one's controlling behavior or propensity for perpetrating IPV increases. This study represents one of the first workplace surveys designed to measure workplace productivity as a function of controlling or violent behavior. Successful results would argue for a more wide-scale testing of the instrument, which could ultimately lead to the development of workplace interventions designed to prevent IPV.

DETAILED DESCRIPTION:
Intimate Partner Violence Intimate partner violence (IPV), which is most often characterized as violence against women, is endemic in our society. Recent data from the National Violence Against Women Survey (NVAWS) suggests that for every 1000 women age 18 and older in the United States, there are 3.2 rape victimizations, 44.2 physical assaults, and 5 stalkings annually. The economic burden of IPV is estimated at $5.8 billion annually, which includes direct medical costs and lost days of work experienced by the victim. A substantial portion of this toll on the economy, at greater than 50%, is borne by our private-sector partners in the form of increased healthcare utilization that is covered by employee health benefits, high employee turnover, decreased productivity, and increased security measures. As businesses become increasingly aware of this burden, more are instituting policies and procedures designed to help victims of IPV in a move to ameliorate the destructive effects of violence on their bottom line.

Recent efforts by the National Center for Injury Prevention and Control=s Division of Violence Prevention have focused prevention efforts targeted towards potential IPV perpetrators rather than victims. The rationale for this new direction in research is the idea that primary prevention that targets potential batterers may ultimately affect the health of women more effectively than targeting secondary/tertiary prevention efforts towards IPV victims. The idea is to stop potential batterers from ever abusing an intimate partner in the first place, rather than empowering a victim of abuse to prevent the violence from continuing. However, there is a paucity of data on the risk and protective factors for IPV perpetration and the economic impact that IPV perpetrators have on the health care and business sectors that would warrant such an investment of scarce public health resources. Until this information is known, developing and evaluating primary prevention programs that target potential abusers is quite challenging, as is our ability to engage our private-sector partners to direct their health promotion resources towards these activities.

Workplace Productivity Employers are increasingly interested in identifying and measuring the relationship between the health issues of their employees and work productivity. Information about this relationship can help guide employers on what types of prevention interventions will be most effective and cost-effective. Performance measures to assess productivity must reflect specific aspects of work output, at a specific point in time, for a specific person. However, only a few modern jobs (e.g., a factory line worker) require workers to perform repetitive tasks that can be easily counted or tracked. Even in industries where employee performance can be tracked objectively, companies often lack reliable systems to capture and review such data. Proxies such as promotions or pay raises also lack the detail necessary to connect a health outcome or behavior with a worker's ability to perform. Without defined business criteria and established metrics to monitor daily output and individual performance, an obvious alternative is asking employees to self-rate their own performance.

Several self-assessment instruments are currently being used in a research setting to estimate work performance and detect the effects of health on performance and productivity (1). Depending upon the health issue(s) under investigation, different instruments may be more or less helpful. In some cases, e.g., measuring the impact of arthritis on productivity, the physical aspect of work might be the most important dimension of productivity to measure. In other cases, questions about "how often" work was affected may be less important than "how much" work was affected. In general, the most important dimensions of work to capture include: physical effort, social interactions, memory or concentration. For example, some jobs involve high risk if a person is fatigued or distracted (bus drivers), others do not. Some jobs require the use of replacement workers (e.g., police or teachers) when a person misses work because of a health issue, others do not. Whatever the occupation, certain aspects of work performance will be affected. Self-assessment tools can be specifically tailored to measure the work impact of controlling behavior on an employee's productivity - as measured by days missed from work - also called absenteeism, and reduced on-the-job productivity - also called presenteeism.

Justification for the current study A major challenge in encouraging the private sector to consider funding workplace promotion and prevention interventions is to provide evidence of returns on investment. One way to do this is by providing evidence that, if not addressed, disease and injury can lead to reductions in individual productivity and overall workplace productivity that can result in substantial losses to the company. To provide this evidence for IPV prevention, this involves measuring productivity in the baseline population and comparing those productivity levels with persons with elevated levels of controlling behavior, violence, or propensity for perpetrating IPV.

Quantifying this relationship is a first step towards understanding the potentially devastating effects that IPV has on our society in general and for the business sector in particular. These data could be instrumental in making the business case for investment in effective and cost effective workplace health promotion interventions that focus on domestic violence perpetrators, in addition to victims, with the ultimate goal of reducing the incidence of IPV in our communities.

Trying to identify people who behave in controlling ways (some of them illegal) towards their intimate partners through a workplace-based anonymous survey do not have implications for the employer in terms of "duty to warn" or other reporting requirements. First, no personal identifiers will be collected through this survey, so it would not be possible to make any reports. We will not have any names, ID numbers, or any other information that would permit reporting a person to the police or referring him or her to treatment. Second, the employer will never see the data. Only the researchers will be able to view the data, which removes the employer from the information loop entirely, much as school administrators are protected when students at their high schools report recent marijuana use on the YRBS. Third, "duty to warn" requirements are applicable when a person has specific knowledge about a crime that is going to occur-not if they have a generalized sense that a person may at some time have engaged in any form of abusive behavior, or even less specifically, that a person has a "propensity for abuse" (which is what this project will collect). This survey will not collect explicit information about criminal abuse perpetration that has occurred in the immediate past, present or immediate future. Fourth, it is essential for victim safety that victims know exactly when they may be at sharply increased risk of harm due to any type of intervention with the perpetrator. Perpetrators may assume the victim is responsible for the report, or blame her for the consequences of the report, and thus may be in more danger because of the third-party report than if no report had been made. Significant work has been done to discourage third-party IPV reporting in the healthcare community for precisely this reason.

The HEALTHY PEOPLE 2010 objectives addressed by this proposal include:

15-32 Reduce the rate of physical assault by current or former intimate partners to 3.6 physical assaults per 1,000 persons aged 12 years and older.

15-35 Reduce the annual rate of rape or attempted rape to 0.7 rapes or attempted rapes per 1,000 persons.

15-36 Reduce sexual assault other than rape to 0.2 sexual assaults other than rape per 1,000 persons aged 12 years and older.

15-37 Reduce physical assaults to 25.5 physical assaults per 1,000 persons aged 12 years and older.

As described previously, violence against women results in substantial morbidity and mortality in our society, with over 50 victimizations occurring annually for every 1000 women over the age of 18. The economic toll is considerable and the private sector, by virtue of subsidizing healthcare insurance and providing employee leave benefits, incurs at least half of the costs associated with IPV. Since employers are in the unique position to offer health promotion and prevention initiatives that can target potential (and confirmed) perpetrators and victims of domestic violence, it is critical for CDC to stimulate these initiatives and to provide evidence-based recommendations where applicable. Stimulating initiatives first requires evidence that domestic abuse affects the employer. While some information is known about how a victim of domestic violence affects the workplace, little is known about how the IPV perpetrator affects the workplace. Targeting research efforts towards the primary prevention of IPV is a newly developing initiative for NCIPC, as is our interest in collaborating with the private sector. This research study provides a unique opportunity to further both of these priorities and to advance our overall mission to reduce the incidence of violence against women in our society.

Overview of the present study The current project involves the pilot testing of an employer-based self-assessment tool to measure productivity. The goals of this research project are 1) to identify the relationship between controlling behavior/propensity for abusiveness and work productivity, 2) to quantify productivity losses for persons with elevated controlling behaviors, and 3) to provide feedback on the research findings to the business community.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be recruited from the Maine Department of Labor (MDOL).

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630
Dates: Start 2004-11; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rothman, ScD, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States